CLINICAL TRIAL: NCT06115785
Title: Evaluation of the Effect of Cognitive Stimulation Therapy on Cognitive Status and Apathy in Olderly People With Mild Cognitive Impairment
Brief Title: Cognitive Stimulation Therapy and Olderly People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ejdane Coskun (Other)
Responsible Party: Sponsor-Investigator, Ejdane Coskun, PhD, Lecturer, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CST
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive stimulation therapy; Mild Cognitive Impairment; Cognitive Status; Apathy
MeSH Terms: conditions — Cognitive Dysfunction; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Stimulation Therapy (Experimental): Cognitive Stimulation Therapy In the 2nd, 3rd, 4th, 6th, 7th and 8th weeks, IPT implementation twice a week, as two themes, for 7 weeks, with each session of 45 minutes.
  Interventions: Behavioral: Cognitive Stimulation Therapy
- CST nonpharmacological intervention (No Intervention): CST nonpharmacological intervention Individuals in the control group will be given two sessions in the 2nd week, and they will continue their daily lives in the following weeks.

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy — Cognitive Stimulation Therapy CST consists of 14 sessions, each session with different themes. The materials used in therapy will differ according to the characteristics of each theme. For example; In the theme of physical games, one of the individuals will be selected by voting, and each individual will be asked to choose a song suitable for the theme and introduce himself/herself to the music accompaniment. Then, a small table game will be prepared with the rackets and ball used for table tennis, and individuals will be able to play a round of table tennis with the researcher and their groupmates. Sessions 10 min. introductory part, 25 min. activity section and in progress10 min. 45 minutes in total, including the ending.
  Other Names: CST nonpharmacological intervention
  Arms: Cognitive Stimulation Therapy

SUMMARY:
The aim of this study is to examine the effect of cognitive stimulation therapy on cognitive status and apathy in elderly individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
This randomized controlled experimental study is planned for 30 October - 25 December 2023, with a total of 60 people (30 in the control group and 30 in the intervention group) at the Elderly Care and Rehabilitation Center. The data of the research were collected from the Literature-Based Personal Information Form, Standardized Mini Mental Test (SMMT), Apathy Assessment Scale. Approval from the Clinical Research Ethics Committee and written permission from the participants were obtained to conduct the study. Individuals in the intervention group started with introduction and in the first week, pre-test administration and CST will be administered twice for 45 minutes.

For the next 7 weeks, it will be carried out for one week, with the introduction and pre-test application for individuals in the control group in the first week. They will continue their daily lives in two sessions for one week and two days. They will continue their lives in the following weeks.

Written informed consent form will be given to all individuals in the study. It will start after information about the measurement tools is given.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* Being literate and speaking Turkish fluently
* Have communication and understanding skills
* Standardized Mini Mental Test result being between 18-23 points
* Having adequate vision and hearing functions for group participation

Exclusion Criteria:

* Presence of any sensory impairment
* Having a physical health problem that may impair group cohesion and integrity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test (SMMT) | up to 9 weeks
  This test consists of 11 items grouped into five subgroups measuring cognitive functions: orientation, recording memory, attention and calculation, recall and language. In SMMT, which is evaluated out of a total of 30 points, one point is given for each correct answer. Although scores of 23/24 for SMMT are considered the limit score for dementia; SMMT score between 18-23 points is considered as mild stage, 10-17 points as moderate stage, and 10 points or less as severe dementia.

SECONDARY OUTCOMES:
Apathy Rating Scale (ARS) | up to 9 weeks
  ARS focuses on the hobbies and pursuits of the individual in his daily life and his enjoyment of them, and measures his loss in these areas.ARS contains a total of 18 items and provides a four-point Likert type measurement. Scores are given between 1 and 4, with 1 representing not at all characteristic and 4 representing very characteristic.The 6th, 10th and 11th items of the scale are in the reverse direction and scoring is done in the reverse direction accordingly.The total score of ARS is found by summing the scores obtained from each of the items and is 18-72.

CONTACTS AND LOCATIONS:
Overall Officials: Ejdane Coşkun, Lect., Principal Investigator — ejdanecoskun@osmaniye.edu.tr
Locations (1):
- Türkiye, Osmaniye, Korkut Ata University, Turkey (Türkiye)

REFERENCES:
- See also: WHO — https://www.who.int
- See also: UCL HomeInternational Cognitive Stimulation Therapy (CST) Centre International Cognitive Stimulation Therapy (CST) Centre — https://www.ucl.ac.uk/international-cognitive-stimulation-therapy/international-cognitive-stimulation-therapy-cst-centre